CLINICAL TRIAL: NCT03365687
Title: Vitamin D In the Prevention of Viral-induced Asthma in Preschoolers: a Randomized Controlled Multicenter Trial (DIVA)
Brief Title: Vitamin D In the Prevention of Viral-induced Asthma in Preschoolers
Acronym: DIVA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Professor Francine Ducharme (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); EURO-PHARM International Canada, Inc. (Other)
Responsible Party: Sponsor-Investigator, Professor Francine Ducharme, Pediatrician, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MP-21-2018-1657
Record Dates: First submitted 2017-12-03; First posted 2017-12-07 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Asthma; Asthma Exacerbations; Preschool Child; Vitamin D; Upper Respiratory Infection; Randomized Controlled Study; Symptoms; Bronchodilator Agents
Keywords: Children; Vitamin D; Respiratory viral infection; Randomized controlled trial; Asthma exacerbations; intervention; functional status; acute care visits; oral corticosteroids; hypercalciuria; hypercalcemia
MeSH Terms: conditions — Asthma; Respiratory Tract Infections; Hypercalciuria; Hypercalcemia | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: This is a randomised, triple-blind, placebo-controlled, parallel-group multicentre trial of vitamin D3 supplementation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The manufacturer, Europharm, will provide the active vitamin D3 and placebo preparations, identical in appearance and taste, in coded latex-free bottles. A web-based randomisation system will allow Site pharmacies to obtain allocated treatment number, prepare the 2 mL bolus in coded syringes and the coded bottles containing the daily dose, and dispense study drugs in masked kits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Active Comparator): Vitamin D supplement (100,000 IU) orally at baseline and at 3.5 months with daily 400 IU vitamin D for 7 months
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Placebo orally at baseline and at 3.5 months with daily placebo during 7 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — 2 mL of 50,000 IU/mL at baseline and at 3.5 months with a daily dose of 1 mL (400 IU/mL) for 7 months
  Other Names: Cholecalciferol
  Arms: Vitamin D
Dietary Supplement: Placebo — 2 mL of placebo at baseline and at 3.5 months with a daily dose of placebo (1 mL) for 7 months
  Arms: Placebo

SUMMARY:
In this 7-month randomized controlled trial, children aged 1 to less than 6 years, with recurrent asthma attacks triggered mostly by colds, will receive a high dose of vitamin D or a placebo every 3.5 months during their usual clinic visit, and a daily supplement of vitamin D or a placebo. This study will test whether children in vitamin D group have less frequent and less severe asthma exacerbations compared with those receiving placebo.The study will also document the safety profile of this strategy.

DETAILED DESCRIPTION:
This is a multicenter triple-blind randomized parallel-group, placebo-controlled trial of vitamin D3 supplementation. Children aged 1-5 (<6) years with physician-diagnosed asthma predominantly triggered by upper respiratory tract infections will be screened for enrolment in paediatric asthma, respiratory or allergy clinics and the ED departments and randomized between Sept 1 to January 31, annually (4 recruitment years) and year around from 2022 onwards.

Using a computer-generated random list, stratified by site, children will be allocated (1:1) using permuted block randomisation method to enhance concealment.

Children will be followed for 7 months, with 3 visits every 3.5 months with repeated urine (for calcium:creatinine ratio) and blood samples. In addition, ten (10) days after each bolus, urine will be sampled for urinary calcium:creatinine ratio. In case of elevated urine calcium:creatinine ratio, a blood sample may be needed primarily for markers of calcium metabolism and exploratory outcomes. Only patients enrolled at CHU Sainte-Justine and Montreal Children's Hospital will receive a systematic home visit 10 days after first bolus for both urine and blood samples. There will be 6 follow-up phone calls, at week 1 and then monthly, to inquire about exacerbations and URTIs, remind parents to complete questionnaires and to collect a nasal swab at each exacerbation and screen for adverse events.

The main outcome is the number of courses of rescue oral corticosteroids (OCS) per child during the study period. Several secondary outcomes will be documented using biological samples and validated questionnaires to ascertain laboratory-confirmed respiratory infections, intensity and severity of exacerbations, mean number of ED visits, parents' functional status during exacerbations, de-intensification of preventive asthma therapy, cost effectiveness, and safety profile.

A sample of 432 children (400+7,5% attrition) per arm will provide 80% power with a two-tailed alpha of 5% to detect a 25% relative reduction in the mean number of exacerbations requiring OCS per child.

An intention-to-treat (ITT) analysis will be carried out with all randomised children.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-5 years
* Physician-diagnosed asthma (as per the 2015 Canadian Position Paper on the diagnosis of preschool asthma)
* ≥1 asthma exacerbation requiring rescue oral corticosteroids (OCS) in the past 6 months or ≥2 in the past 12 months; or from the pandemic (2020) onwards, ≥1 asthma exacerbation requiring rescue oral corticosteroids (OCS) in the past 12 months (as documented by pharmacy/medical records)
* ≥4 upper respiratory tract infections (URTIs) in the past 12 months (as per parental report); or from the pandemic (2020) onwards, ≥ 2 URTIs in past 12 months
* URTIs as the main asthma trigger (as per parental report)

Exclusion Criteria:

* Intake > 400 IU/day of vitamin D3 supplements or fish oil in the past 3 months
* Intention to use > 400 IU/day of vitamin D3 supplements or fish oil in the fall and winter
* Extreme prematurity (< 28 week gestation)
* No vitamin D supplementation (if breast-fed in the last 6 months)
* Vitamin D restrictive diets, that is, minimal intake of vitamin D fortified milk (<250 mL/day for 1-3 years or <375 mL/day for 4-6 years AND no other (or <200 IU/day) vitamin D supplement
* Recent immigrants from regions at high risk of rickets (in the past 12 months)
* Recent refugees (in the past 12 months)
* Undernourished children
* Other chronic respiratory disease (e.g. Cystic fibrosis, Bronchopulmonary dysplasia) or chronic kidney, gastrointestinal, endocrinological or cardiac diseases, or sickle cell anemia
* History of bone disorder disease (e.g. rickets, osteomalacia)
* Intake of oral anti-epileptic, diuretic or anti-fungal medications
* Anticipated difficulty with follow-up or with adherence to the intervention or the procedures

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 323 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of asthma exacerbations per child treated with rescue oral corticosteroids | 7 months
  Group difference in the mean number of exacerbations treated with rescue oral corticosteroids/child

SECONDARY OUTCOMES:
Laboratory-confirmed respiratory infections | 7 months
  Group difference in (i) mean number of laboratory-confirmed respiratory infections per child and (ii) distribution of viruses during colds and/or asthma exacerbations
Mean number of ED visits and hospital admissions for asthma exacerbations | 7 months
  Group difference in mean number of ED visits and hospital admissions for asthma exacerbations per child
De-intensification of preventive asthma therapy | 3.5 and 7 months
  Group difference in proportion of children with de-intensification of preventive asthma therapy
Duration of asthma symptoms during asthma exacerbations | 7 months
  Group difference in the mean duration of symptoms during asthma exacerbations per child (i) documented in writing on the validated 'Asthma Flare-up Diary for Young Children' and (ii) reported verbally by parents,
Duration of B2-agonist use during asthma exacerbations | 7 months
  Group difference in the mean duration of B2-agonist use during asthma exacerbations per child (i) documented in writing on the validated 'Asthma Flare-up Diary for Young Children' and (ii) reported verbally by parents,
Severity of asthma symptoms during asthma exacerbations | 7 months
  Group difference in the severity of symptoms during asthma exacerbations per child documented on the 'Asthma Flare-up Diary for Young Children'
Intensity of use of rescue β2-agonists during asthma exacerbations | 7 months
  Group difference in the mean cumulative use of rescue β2-agonists per child during exacerbations documented on the validated 'Asthma Flare-up Diary for Young Children'
Parents' functional status during asthma exacerbations | 7 months
  Group difference in the mean parents' functional status during asthma exacerbations per child as documented on the validated 'Effect of a child's asthma flare-up on parents questionnaire'
Number of parental workdays lost | 7 months
  Group difference in the cumulative number of days of work or regular planned activities missed by parents to care for their child during asthma exacerbations
Parental productivity | 7 months
  Group difference in the extent to which parents were able to perform their work or regular planned activities during their child's acute asthma exacerbation (%)
Intervention cost-effectiveness | 7 months
  Cost of intervention vs. cost (family expenses and health care) of exacerbations

OTHER OUTCOMES:
Hypercalcemia | 7 months
  Group difference in the proportion of children with clinically significant hypercalcemia (>2.63 mmol/L)
Hypercalciuria | 7 months
  Group difference in the proportion of children with ≥1 occurrence of hypercalciuria (urinary calcium: creatinine ratio >1.38 mmol/mmol for children aged 1-<2 years, or >1.1 mmol/mmol for children aged 2-<5 years, or >0.77 mmol/mmol for children aged ≥5 years)
Elevated serum 25-hydroxyvitamin D | 7 months
  Group difference in the proportion of children with ≥1 occurrence of elevated serum 25OHD (greater than 250 nmol/L)
Adverse Health Events | 7 months
  Group difference in the number and distribution of adverse health events
Serious Adverse Health Events | 7 months
  Group difference in the number of serious adverse health events
Gene expression | 3.5 months
  Group difference in the change in gene expression levels (between baseline and 3.5 months) in peripheral blood mononuclear cells (PBMC) in a subset of patients

CONTACTS AND LOCATIONS:
Overall Officials: Francine M Ducharme, MD, Principal Investigator — Study Principal Investigator
Locations (9):
- Canada (9):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Children's Hospital of London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - CHU Sainte Justine, Montreal, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
  - CHU de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: approximatively 18 months from datalock (Dec 2026)
Access Criteria: to be determined

REFERENCES:
- [Background] Jensen ME, Ducharme FM, Alos N, Mailhot G, Masse B, White JH, Sadatsafavi M, Khamessan A, Tse SM, Alizadehfar R, Bock DE, Daigneault P, Lemire C, Yang C, Radhakrishnan D. Vitamin D in the prevention of exacerbations of asthma in preschoolers (DIVA): protocol for a multicentre randomised placebo-controlled triple-blind trial. BMJ Open. 2019 Dec 30;9(12):e033075. doi: 10.1136/bmjopen-2019-033075. PMID 31892662

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-05-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT03365687/SAP_000.pdf